CLINICAL TRIAL: NCT03437525
Title: Peer Support in Diabetes Management - Insulin Peer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Asian Center for Health Education (Other); Shanghai Municipal Commission of Health and Family Planning (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Weiping Jia, Professor, President of Shanghai 6th People's Hospital, Director of Shanghai Institute of Diabetes, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-73
Record Dates: First submitted 2018-01-24; First posted 2018-02-19 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Diabetes; Self-Management; Primary Care; Community Health Center; Peer Support; Group Support; Integrated Care; Insulin; China; Urban
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study uses a cluster randomized controlled trial design with one experimental condition and one control condition. Ten community health centers (CHC) will be randomized to either the experimental or control condition. The five CHCs in the experimental group will deliver the peer support intervention for 12 months and the five CHCs in the control group will deliver usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Support Intervention (Experimental): The experimental group will receive the peer support intervention for 12 months.
  Interventions: Behavioral: Peer Support
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Peer Support — The intervention involves monthly education/support groups co-led by a CHC doctor / nurse and peer coaches. These meetings will begin with a general discussion about participants' previous month, what they had been doing, any special events etc. Meetings will devote time to identifying goals and specific plans for reaching them, rehearsal and/or discussion of specific behaviors to execute plans and ways in which the group members can be helpful to each other. This will be organized around a Diabetes Action Plan. Peer coaches will provide education and support for insulin therapy to help reduce barriers around insulin use. Peer coaches will also organize activities to promote healthy lifestyles, such as walking groups, to promote informal contacts among peer supporters and participants.
  Arms: Peer Support Intervention

SUMMARY:
This project will develop a combined model of the Shanghai Integration Model and peer support for diabetes self-management with a special focus on appropriate insulin use.

DETAILED DESCRIPTION:
The development of contemporary diabetes care offers new hope for long and satisfying lives of those with the disease, but also provides increased challenges for integration across the many dimensions of care (varied medications in addition to insulin, specialty services, diet, physical activity, stress management, etc.) and across the many who contribute to care (specialists, primary care providers, nurses, dietitians and patient educators, family members, friends, worksites). The Shanghai Integration Model (SIM) has made great strides to integrating specialty/hospital care with primary/community care. The addition of peer support can enhance patient engagement within that integrated care. Peer support can also integrate care with the daily behaviors and patterns that optimal diabetes management requires and with the family members and others in individuals' daily lives who can support diabetes management.

The "Insulin Peer Support" project is a sub-project of "Peer Support in Diabetes Care", with special focus on appropriate insulin use in the community, to help overcome barriers in insulin treatment and improve treatment compliance. This project will develop a peer support model for diabetes management in Chinese patients undergoing insulin treatment and evaluate its effectiveness in a randomized controlled trial of 10 CHCs in Shanghai.

The project is a collaboration among the Shanghai Sixth People's Hospital, Shanghai Jiao Tong University, the Shanghai Diabetes Institute,the Shanghai Municipal Commission of Health and Family Planning, the Shanghai Centers for Disease Control, and, at the University of North Carolina-Chapel Hill, Peers for Progress, widely recognized for its leadership in promoting peer support in health care and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Has type 2 diabetes
* Receiving treatment at participating community health center
* Currently using insulin or prescribed insulin but not currently using insulin

Exclusion Criteria:

* Severe mental illness (severe depression, schizophrenia, bipolar disorder, obsessive compulsive disorder, panic disorder, PTSD, borderline personality disorder, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 6 and 12 months | Baseline, 6 months, 12 months
  HbA1c (%)

SECONDARY OUTCOMES:
Change from Baseline Fasting Blood Glucose at 6 and 12 months | Baseline, 6 months, 12 months
  FPG (mmol/L)
Change from Baseline Blood Pressure at 6 and 12 months | Baseline, 6 months, 12 months
  SBP and DBP (mmHg)
Change from Baseline BMI at 6 and 12 months | Baseline, 6 months, 12 months
  Height (cm) and weight (kg)
Change from Baseline Blood Lipids at 6 and 12 months | Baseline, 6 months, 12 months
  Total cholesterol, triglycerides, HDL, LDL (mmol/L)
Change from Baseline Hemoglobin at 6 and 12 months | Baseline, 6 months, 12 months
  Hemoglobin (g/L)
Change from Baseline Red Blood Cell Count at 6 and 12 months | Baseline, 6 months, 12 months
  Red blood cell count (10^12/L)
Change from Baseline Mean Corpuscular Volume at 6 and 12 months | Baseline, 6 months, 12 months
  Mean Corpuscular Volume (fL)
Change from Baseline Mean Corpuscular Hemoglobin at 6 and 12 months | Baseline, 6 months, 12 months
  Mean Corpuscular Hemoglobin (pg)
Change from Baseline Liver Functioning at 6 and 12 months | Baseline, 6 months, 12 months
  ALT (U/L), AST (U/L), Alkaline phosphatase (U/L), r-GT (U/L)
Change from Baseline Bilirubin at 6 and 12 months | Baseline, 6 months, 12 months
  Total bilirubin (µmol/L), Direct bilirubin (µmol/L)
Change from Baseline Blood Urea at 6 and 12 months | Baseline, 6 months, 12 months
  Blood urea (mmol/L)
Change from Baseline Serum Creatinine at 6 and 12 months | Baseline, 6 months, 12 months
  Serum creatinine (µmol/L)
Change from Baseline Uric Acid at 6 and 12 months | Baseline, 6 months, 12 months
  Uric acid (µmol/L)
Change from Baseline Urine Albumin/Creatinine Ratio at 6 and 12 months | Baseline, 6 months, 12 months
  Albumin (mg/L), Creatinine (mmol/L)
Change in Insulin Functioning at 6 and 12 months | 6 months, 12 months
  Insulin (pmol/L)
Change in C-peptides at 6 and 12 months | 6 months, 12 months
  C-peptide (nmol/L)
Change from Baseline Diabetes Self Care Behaviors at 6 and 12 months | Baseline, 6 months, 12 months
  9 items from Summary of Diabetes Self Care Activities and Behavioral Risk Factor Surveillance System. Items 1-7 measure diabetes self care activities during the previous 7 days. Items 1, 2, 4-7 are assessed on a scale of 0 to 7 days. Item 3 is assessed on scale of 1-4, where 1 represents very low levels of daily activity and 4 represents very high levels of daily activity. Items 8 and 9 are yes/no questions that measure cigarette intake over the past 7 and 30 days.
Change from Baseline Medication Adherence at 6 and 12 months | Baseline, 6 months, 12 months
  Morisky 4-item adherence scale. Four yes/no questions about medication adherence in which yes responses are less favorable. Yes responses are coded as 0, No responses are coded as 1, and scores are summed. A total score of 0 is the lowest level of medication adherence and 4 is the highest level of medication adherence.
Change from Baseline General Quality of Life at 6 and 12 months | Baseline, 6 months, 12 months
  6-item EQ-5D, a standardized instrument for measuring generic health status. The respondents are asked to choose one of the statements which best describes their health status on the surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Item 6 is the visual analogue scale, in which respondents are asked to mark their health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100, where 0 corresponds to "the worst health you can imagine", and 100 corresponds to "the best health you can imagine"
Change from Baseline Diabetes Quality of Life at 6 and 12 months | Baseline, 6 months, 12 months
  4-item Diabetes Distress Scale, an abbreviated version of the 17-item Diabetes Distress Scale. The respondents are asked to respond to which degree each of the items has bothered them in the past month on a 6-point scale (1-6), where 1 is not a brother and 6 is very bothersome. Scores are summed and divided by 4 to calculate the mean. Mean scores of 3 or higher (moderate distress) are considered worthy of clinical attention.
Change from Baseline Depression at 6 and 12 months | Baseline, 6 months, 12 months
  8-item Patient Health Questionnaire (PHQ), the PHQ-9 minus the last question on suicidal thoughts. The PHQ is a standard instrument used in primary care settings to screen for the presence and severity of depression. The respondents are asked how often they have been bothered by each of the 8 items in the past 2 weeks on a 4 point scale (0-3), where 0 is "not all" and 3 is "nearly every day". The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Change in Community Support for Diabetes at 6 and 12 months | 6 months, 12 months
  Novel 9-item questionnaire that assesses the degree to which respondents receive community support (other than family) for their diabetes. Items 1-8 are scored from on a scale of 1-5, where 1 is "not at all" and 5 is "completely". Item 9 asks for the relationship of the person / people to the respondent.
Change in Healthcare Utilization at 6 and 12 months | 6 months, 12 months
  Novel 6-item questionnaire that assesses patterns of healthcare and program utilization. Item 1 asks respondents the last time they saw a community health center doctor or nurse for their diabetes. Possible responses are "Within the last 2 weeks", "Within the last month", "Within the last 2 months", "Between 2-4 months ago", and "More than 4 months ago". Items 2-6 ask respondents to recall how many times they accessed healthcare services (peer support, primary care, outpatient hospital care, overnight hospital stays) in the past 3 months. Possible responses are "0", "1-2", "3-5", and "5+".
Change from Baseline Insulin Attitudes at 6 and 12 months | Baseline, 6 months, 12 months
  13-item Chinese Attitudes to Starting Insulin Questionnaire (Ch-ASIQ). Four subscales consisting of 'Self-image and stigmatization' (3 items); 'Factors promoting self-efficacy (5 items); 'Fear of pain or needles' (3 items); and 'Time and family support' (2 items). Responses are scored using a 4-point Likert scale (Totally disagree = 1, Totally Agree = 4). Individual scale scores are calculated by summing the item responses. For the subscales 'Factors promoting self-efficacy' and 'Time and family support', higher scores indicate more positive attitudes towards the use of insulin. For the subscales 'Self-image and stigmatization' and 'Fear of pain or needles' a higher score indicates a more negative attitude towards insulin initiation. The weighted sum of all four scale scores, converting two positively coded scales to negatively coded scales, calculates the overall score with higher scores indicating more negative attitude to starting insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, PhD, Principal Investigator — Shanghai 6th People's Hospital; Edwin B Fisher, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (11):
- China (11):
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - An Ting Community Health Center, Shanghai, Shanghai Municipality
  - Cao He Jing Community Health Center, Shanghai, Shanghai Municipality
  - Cao Yang Community Health Center, Shanghai, Shanghai Municipality
  - Hong Mei Community Health Center, Shanghai, Shanghai Municipality
  - Kang Jian Community Health Center, Shanghai, Shanghai Municipality
  - Long Hua Community Health Center, Shanghai, Shanghai Municipality
  - Nan Jing Xi Road Community Health Center, Shanghai, Shanghai Municipality
  - Tao Pu Community Health Center, Shanghai, Shanghai Municipality
  - Tian Lin Community Health Center, Shanghai, Shanghai Municipality
  - Zhen Ru Community Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher EB, Boothroyd RI, Coufal MM, Baumann LC, Mbanya JC, Rotheram-Borus MJ, Sanguanprasit B, Tanasugarn C. Peer support for self-management of diabetes improved outcomes in international settings. Health Aff (Millwood). 2012 Jan;31(1):130-9. doi: 10.1377/hlthaff.2011.0914. PMID 22232103
- [Background] Zhong X, Wang Z, Fisher EB, Tanasugarn C. Peer Support for Diabetes Management in Primary Care and Community Settings in Anhui Province, China. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S50-8. doi: 10.1370/afm.1799. PMID 26304972
- [Background] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960